CLINICAL TRIAL: NCT03766958
Title: An Observational Registry Study to Evaluate the Performance of the BDX-XL2 Test
Brief Title: A Registry to Evaluate the Performance of the BDX-XL2 Test
Acronym: ORACLE
Status: Completed | Type: Observational
Sponsor: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BDX-CD-002
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Nodule Solitary Pulmonary; NSCLC
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Registry Patients With Nodify Lung Results: Patients providing consent to have data collected to observe how Nodify Lung results were used in the clinical management of their lung nodules.
- Contemporaneous Group Without Nodify Lung: Contemporaneous group who did not have Nodify Lung test results for use in the clinical management of their lung nodules.

SUMMARY:
The purpose of the ORACLE Registry is to demonstrate clinical utility of the BDX-XL2 test; specifically, the potential to reduce unnecessary invasive procedures, such as biopsies and surgeries, on benign lung nodules while not significantly increasing the number of malignant lung nodules routed to CT surveillance. Clinical data will be collected from participating patients to evaluate the impact of the BDX-XL2 test when used in the clinical management of recently identified lung nodules assessed to have a low to moderate risk of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided informed consent to participate in the registry and agrees to comply with all protocol requirements.
2. Patient meets the criteria for the intended use population of Nodify Lung testing:

   * Patient is > 40 years of age at the time of the discovery of the lung nodule of concern.
   * The maximal dimension of the patient's lung nodule of concern is > 8mm and < 30mm.
   * The pre-test risk of cancer as determined by the Mayo risk prediction algorithm is 65% or less.
3. The first CT scan identifying the lung nodule of concern was performed within 60 days of patient enrollment in the registry.

Exclusion Criteria:

1. Nodule work-up before the time of patient enrollment indicating any attempted or completed biopsy procedure after the first CT scan identifying the lung nodule of concern.
2. High risk per physician assessment (i.e. > 65% by physician pCA)
3. Current diagnosis of any active cancer.
4. Prior diagnosis of lung cancer.
5. Prior diagnosis of any cancer within 5 years of lung nodule detection, except for non-melanomatous skin cancer.
6. Concurrent participation in any unrelated clinical trial that may impact or alter the management of the patient's nodule of concern.
7. Any illness or factor that will prevent compliance with follow-up as recommended.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified from the patient populations of participating pulmonary medicine practices.
Sampling Method: Non-Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Statistically significant change in the proportion of benign lung nodules managed by Nodify Lung experiencing invasive procedures. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steve Springmeyer, Principal Investigator — Biodesix, Inc.; Michael Pritchett, DO, Principal Investigator — Pinehurst Medical Clinic
Locations (15):
- United States (15):
  - Banner Health, Sun City, Arizona
  - Amicis Research Center, Northridge, California
  - Pueblo Pulmonary Associates, Pueblo, Colorado
  - Stamford Health, Stamford, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Nevada, Las Vegas, Las Vegas, Nevada
  - East Carolina University, Greenville, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Clinical Research Associates of Central PA/Penn Highlands Hospital, DuBois, Pennsylvania
  - Peacehealth, Bellingham, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Pritchett MA, Sigal B, Bowling MR, Kurman JS, Pitcher T, Springmeyer SC; ORACLE Study Investigators. Assessing a biomarker's ability to reduce invasive procedures in patients with benign lung nodules: Results from the ORACLE study. PLoS One. 2023 Jul 11;18(7):e0287409. doi: 10.1371/journal.pone.0287409. eCollection 2023. PMID 37432960